CLINICAL TRIAL: NCT04411628
Title: A Randomized, Placebo-Controlled, Double-Blind, Sponsor Unblinded, Single Ascending Dose, Phase 1 First in Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous LY3819253 in Participants Hospitalized for COVID-19
Brief Title: A Study of LY3819253 (LY-CoV555) in Participants Hospitalized for COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AbCellera Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17823; J2W-MC-PYAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — bamlanivimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3819253 (Experimental): Participants received single doses of 700 milligrams (mg), 2800 mg or 7000 mg LY3819253 administered as intravenous infusion.
  Interventions: Drug: LY3819253
- Placebo (Placebo Comparator): Participants received single dose of Placebo as intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3819253 — Administered IV.
  Other Names: LY-CoV555; Bamlanivimab
  Arms: LY3819253
Drug: Placebo — Administered IV.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and tolerability of LY3819253 when it is given by injection into a vein to participants hospitalized with COVID-19. Blood tests will be done to check how much LY3819253 is in the bloodstream and how long the body takes to eliminate it. Participation could last about 8 weeks and may include up to 15 visits in the hospital or the home.

ELIGIBILITY:
Inclusion Criteria:

* Are hospitalized or in the process of being admitted to hospital and have an initial laboratory determination of current COVID-19 infection less than or equal to (≤)72 hours prior to randomization
* Are men or non-pregnant women
* Women of childbearing potential must agree to use at least one highly effective form of contraception for the entirety of the study
* Agree to the collection of nasopharyngeal swabs and venous blood

Exclusion Criteria:

* Require mechanical ventilation or anticipated impending need for mechanical ventilation
* Received convalescent COVID-19 plasma treatment prior to enrollment
* Were resident in a nursing home or long-term care facility immediately prior to current hospitalization
* Suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking investigational product
* Have an oxygen saturation (SpO2) less than (<)88 percent (%) while breathing room air at rest at randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (11):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Veterans Affairs Medical Center San Diego, San Diego, California
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Alexandria Center for Life - NYC/ NYCEDC, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Unified Research Enterprise Brody School of Medicine at ECU, Greenville, North Carolina
  - Temple Univ School of Med, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Nathan R, Shawa I, De La Torre I, Pustizzi JM, Haustrup N, Patel DR, Huhn G. A Narrative Review of the Clinical Practicalities of Bamlanivimab and Etesevimab Antibody Therapies for SARS-CoV-2. Infect Dis Ther. 2021 Dec;10(4):1933-1947. doi: 10.1007/s40121-021-00515-6. Epub 2021 Aug 10. PMID 34374951
- See also: A Study of LY3819253 (LY-CoV555) in Participants Hospitalized for COVID-19 — https://trials.lillytrialguide.com/en-US/trial/3B9kHya2iCF9SHumC5PLKk

RESULTS

PARTICIPANT FLOW:
Groups:
- 700 mg LY3819253 IV: Participants received single dose of 700 milligrams (mg) LY3819253 administered as intravenous infusion.
- 2800 mg LY3819253 IV: Participants received single dose of 2800 mg LY3819253 administered as intravenous infusion.
- 7000 mg LY3819253 IV: Participants received single dose of 7000 mg LY3819253 administered as intravenous infusion.
Period: Overall Study
Arm/Group | Placebo | 700 mg LY3819253 IV | 2800 mg LY3819253 IV | 7000 mg LY3819253 IV
Started | 7 | 6 | 7 | 6
Received at Least 1 Dose of Study Drug | 6 | 6 | 6 | 6
Completed | 6 | 4 | 5 | 6
Not Completed | 1 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 700 mg LY3819253 IV | 2800 mg LY3819253 IV | 7000 mg LY3819253 IV | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.2 (8.6) | 57.2 (6.8) | 48.5 (12.1) | 66.7 (6.7) | 53.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 1 | 7
  Male | 4 | 4 | 4 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 3 | 3 | 15
  Not Hispanic or Latino | 1 | 2 | 3 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 5 | 4 | 5 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is any adverse event that results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. The number of participants with 1 or more SAEs considered by the investigator to be related to study drug administration is reported. A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, were reported in the Reported Adverse Events module.
Time Frame: Baseline through Day 60
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | 700 mg LY3819253 IV | 2800 mg LY3819253 IV | 7000 mg LY3819253 IV
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Mean Concentration of LY3819253 on Day 29
Description: Pharmacokinetics (PK): Mean Concentration of LY3819253 on Day 29.
Time Frame: Day 29
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | 700 mg LY3819253 IV | 2800 mg LY3819253 IV | 7000 mg LY3819253 IV
Number analyzed (Participants) | 4 | 5 | 6
microgram per milliliter (µg/mL) | 28.2 (75) | 59.4 (37) | 261 (50)

3. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline to Day 29 in Viral Load
Description: Pharmacodynamics (PD): Change from Baseline to Day 29 in Viral Load.
Time Frame: Baseline, Day 29
Population: All randomized participants who received at least one dose of study drug and had baseline, post baseline data for viral load.
Measure: Mean (Standard Deviation); unit: log10 (Copies/mL)
Arm/Group | Placebo | 700 mg LY3819253 IV | 2800 mg LY3819253 IV | 7000 mg LY3819253 IV
Number analyzed (Participants) | 5 | 4 | 5 | 5
log10 (Copies/mL) | 10.476 (7.117) | 10.923 (10.036) | 16.956 (10.388) | 15.726 (5.723)

4. Secondary Outcome: Pharmacodynamics (PD): SARS-CoV-2 Viral Load AUC
Description: The SARS-CoV-2 viral load was derived from the cycle time (CT) values using a polymerase chain reaction (PCR) assay. Higher CT values indicate a lower viral load.
Time Frame: Day 1 pre-dose, Days 3, 7, 11, 15, 22, 29 post dose
Population: All randomized participants who received at least one dose of study drug and had data for SARS-CoV-2 viral load AUC.
Measure: Mean (Standard Deviation); unit: Cycles*day
Arm/Group | Placebo | 700 mg LY3819253 IV | 2800 mg LY3819253 IV | 7000 mg LY3819253 IV
Number analyzed (Participants) | 5 | 4 | 5 | 5
Cycles*day | 48.865 (28.020) | 44.858 (40.027) | 60.818 (24.266) | 69.528 (39.336)

5. Secondary Outcome: Pharmacodynamics (PD): Time to SARS-CoV-2 Clearance
Description: Pharmacodynamics (PD): Time to SARS-CoV-2 clearance.
Time Frame: Day 1 pre-dose, Days 3, 7, 11, 15, 22, 29 post dose
Population: All randomized participants who received at least one dose of study drug and had data for SARS-CoV-2 clearance.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | 700 mg LY3819253 IV | 2800 mg LY3819253 IV | 7000 mg LY3819253 IV
Number analyzed (Participants) | 2 | 3 | 2 | 3
Days | NA (NA) — Not calculated as participant number is small. | 7.7 (7.0) | NA (NA) — Not calculated as participant number is small. | 15.7 (11.2)

ADVERSE EVENTS:
Time Frame: Baseline through day 60
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | 700 mg LY3819253 IV | 2800 mg LY3819253 IV | 7000 mg LY3819253 IV
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6 | 5/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | 700 mg LY3819253 IV (N=6) | 2800 mg LY3819253 IV (N=6) | 7000 mg LY3819253 IV (N=6)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT04411628/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT04411628/SAP_001.pdf